CLINICAL TRIAL: NCT01449903
Title: Core Build-up Materials: a Randomized Clinical Study
Brief Title: Survival of Different Core Build-up Materials
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Brigitte Ohlmann, PD Dr. med. dent. Brigitte Ohlmann, Heidelberg University
Other Study IDs: Proth-003
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Dental Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rebilda DC
- Clearfil Core DC / Plus
- Multicore Flow

SUMMARY:
The purpose of this study is to compare three different core build-up materials for dental use. The study hypothesis is that there is no differences in survival rate of the different core build-ups.

DETAILED DESCRIPTION:
Core build-ups replace dental structures which are decayed through caries or tooth fractures. Often there are necessary before insertion of dental restorations. In clinical practice, there are two main material groups: glass ionomer cements and composites. Because of there good physical properties the composite materials claimed to fulfill the expected criteria of core build-ups. However, some of these composite core build-ups get lost before insertion of definite prosthetic restorations. The current prospective, randomized controlled study should investigate the survival rate of three different composite materials: "Rebilda DC", "Clearfil Core DC / Plus" and "Multicore Flow". The statistical analysis will performed with logistic regression performed by the institute of institute of Medical Biometry and Informatics, university of heidelberg. The study hypothesis is that there is no differences in the survival rate.

ELIGIBILITY:
Inclusion Criteria:

* patients need a single crown or fixed dental prostheses
* patients are able to signed inform consent form, more than 18 years,

Exclusion Criteria:

* no pregnant women
* insufficient oral hygiene

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the department of porsthodontics, university of heidelberg
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rammelsberg, Prof. Dr., Principal Investigator — Heidelberg University
Locations (1):
- Department of prosthodontics, university of heidelberg, Heidelberg, Germany